CLINICAL TRIAL: NCT00848640
Title: Multi-center,Middle East, Phase-II Study, Non-comparative, of the RAF-Kinase Inhibitor Sorafenib in Patients With Advanced Renal Cell Carcinoma to Evaluate The Efficacy and Tolerability of the Drug
Brief Title: Study of Sorafenib in Patients With Advanced Renal Cell Carcinoma
Acronym: MERITS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Egyptian Foundation For Cancer Research (Other)
Responsible Party: Hussein Khaled, MD, Egyptian Foundation For Cancer Research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12594
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2009-09

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib (Experimental)
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — 400 mg twice daily

SUMMARY:
The purpose study is to evaluate the efficacy and safety of Sorafenib as first line treatment for patients - unsuitable for another approved first line therapy - with advanced RCC in the Middle East Region.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must provide written informed consent prior to receiving Sorafenib.
2. The male or female patient must be at least 18 years of age.
3. The patient must have pathologically proven advanced Renal Cell Carcinoma.
4. Only patients with measurable disease (According to RECIST) at baseline should be included in protocol where Disease Control Rate (DCR) is the primary endpoint.
5. The patient requires Sorafenib as First line therapy as the patient is unsuitable for another approved first line therapy for advanced RCC.
6. The patient must be, in the Investigator's opinion, reasonably likely to benefit from treatment with Sorafenib as a single agent.
7. The patient must have an Eastern Cooperative Oncology Group performance status of 0 - 2.
8. The patient will not require other systemic anti-cancer chemotherapy, immunotherapy or hormonal therapy, except for bisphosphonates while taking Sorafenib.
9. Both male and female patients must use adequate barrier birth control methods during their participation in the protocol. The birth control methods must be used for 4 weeks for female patients and for 3 months for male patients after discontinuation of treatment with Sorafenib.
10. For patients, who have had major surgery, the wound must be completely healed prior to receiving Sorafenib treatment (4 weeks).
11. The patient must have within normal Renal & Hepatic function.
12. The patient must have within normal CBC.

Exclusion Criteria:

1. Patients who are currently enrolled in or have previously participated in any other Sorafenib trial.
2. Suitable or received any other systemic therapy for treatment RCC (IL-2, INF)
3. Patients who have a life expectancy of less than 2 months.
4. Patients with metastatic brain or meningeal tumours.
5. Patients are excluded who require any of the following:

   * Investigational drug therapy during the treatment with Sorafenib or within 30 days prior to their first dose of Sorafenib.
   * Concomitant Rifampicin.
6. Non-measurable disease according to RECIST.
7. Concomitant St. John's Wort (Hypericum perforatum).
8. Warfarin (or similar medication) is allowed.
9. Women who are pregnant or breast-feeding. Women of childbearing potential must have a negative pregnancy test performed within seven days of the start of study drug (please note that no laboratory data are collected in this study).
10. Patients with congestive heart failure greater than NYHA functional class II (symptomatic during ordinary activity)
11. Patients with cardiac arrhythmias greater than Grade 1 NCI CTCAE, Version 3.0 (conduction abnormality and supraventricular arrhythmia present but patient is asymptomatic; intervention not indicated, palpitations present and QTc > 0.45 - 0.47 second).
12. Patients with active coronary artery disease or ischemia.
13. Patients with Child-Pugh class C hepatic impairment.
14. Patients with severe renal impairment (calculated creatinine clearance of < 30 ml/min) or who require dialysis.
15. Patients with active uncontrolled hypertension.
16. Patients with recent or active bleeding diathesis.
17. Patients with any medical condition which could jeopardize their safety while taking an investigational drug.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
evaluate the efficacy by evaluating the disease control rate (DCR) and safety of Sorafenib for first line patients unsuitable for another approved first line therapy with advanced RCC in the Middle East region. | Disease Control Rate (DCR) defined as either CR, PR or SD for at least 8 weeks

SECONDARY OUTCOMES:
Quality of life of patient with RCC and Progression Free Survival | One year

CONTACTS AND LOCATIONS:
Overall Officials: Hussein M. Khaled, MD, Principal Investigator — Egyptian Foundation For Cancer Research
Locations (1):
- Egyptian Foundation For Cancer Research, Cairo, Egypt